CLINICAL TRIAL: NCT05103709
Title: Effect of Multiple Micronutrient Fortified Bread Consumption on Iron Deficiency Anemia in Women of Reproductive Age: A Randomized Controlled Trial
Brief Title: Effect of Multiple Micronutrient Fortified Bread Consumption on Iron Deficiency Anemia in Women of Reproductive Age
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SIDISI 204220
Record Dates: First submitted 2021-10-25; First posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-07

CONDITIONS: Iron Deficiency Anemia
Keywords: iron deficiency anemia; hemoglobin; iron status; hematological parameters
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Food, Fortified

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Masking will be mixed. Since the third arm will not receive product of any kind it is not possible to mask the volunteers assigned to this group. The packaging of the products will be neutral to blind the volunteers in the groups that will receive products. The investigators will be blinded to randomization at all times.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MULTI-FORTIFIED (Experimental): The product to be evaluated is bread made from wheat flour fortified according to Peruvian national standards [Riboflavin (0.18 mg), niacin (2.25 mg), thiamine (0.18 mg), folic acid (60ug), iron (4.2 mg)] and a previtamin mix [Vitamin A (240 ug), Vitamin b12 (0.72 ug), zinc (5.25 mg) per daily serving]. Participants will receive 2 slices of bread a day for 120 days. It is supplied by Panificadora Bimbo del Peru S.A.
  Interventions: Other: MULTI-FORTIFIED
- FORTIFIED (Active Comparator): The active comparator is bread fortified according to Peruvian national standards [Riboflavin (0.18 mg), niacin (2.25 mg), thiamine (0.18 mg), folic acid (60ug), iron (4.2 mg)]. Participants will receive 2 slices of bread a day for 120 days. It is supplied by Panificadora Bimbo del Peru S.A.
  Interventions: Other: FORTIFIED
- CONTROL (No Intervention): The control group will be followed for 120 days. No product will be provided.

INTERVENTIONS:
Other: MULTI-FORTIFIED — Treatment with multifortified bread for 120 days
  Arms: MULTI-FORTIFIED
Other: FORTIFIED — Treatment with standard bread, fortified according to current Peruvian guidelines for 120 days
  Arms: FORTIFIED

SUMMARY:
The project aims to assess if consuming two slices of multi-fortified bread daily for 120 days is effective in reducing iron deficiency anemia in women of reproductive age through a three-arm randomized trial.

DETAILED DESCRIPTION:
Iron deficiency anemia (IDA) continues to be a public health priority in Peru and the world. The prevalence of the condition is high in women of reproductive age regardless of geographic area and socioeconomic status. Fortification of staple foods is recognized as a cost-effective strategy to reverse iron deficiency. In Peru, iron fortification of wheat flour and derived products is mandatory, but to date its effect on the IDA has not been evaluated. In recent years, evidence has been generated on the positive effect of zinc, vitamin A and vitamin B12 supplementation on hemoglobin (Hb) levels. This project is a three-arm randomized clinical trial that seeks to evaluate the effect of consuming two slices of bread fortified with a multivitamin premix (iron, folic acid, vitamin A, vitamin B12 and zinc) daily on iron deficiency anemia in non-pregnant women of reproductive age. As a control, one group will receive standard bread fortified according to Peruvian legislation and a third group will not receive treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ferritin levels < 13 ng/ml,
* Hemoglobin levels between 8 g/dL and 11.9 g/dL,
* No plans to move during the duration of the study,
* Commitment not to become pregnant during the duration of the study,
* Signed informed consent.

Exclusion Criteria:

* Pregnancy,
* Amenorrhea not related to pregnancy,
* Breastfeeding,
* Chronic diseases (active TB, HIV, cancer, asthma, liver disease, coronary heart disease, chronic renal disease),
* Hemoglobin levels < 8 g/dL,
* Bleeding in the 3 months prior to recruitment,
* Smoking,
* Inability to sign informed consent,
* Consumption of nutritional supplements.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 351 (Estimated)
Dates: Start 2021-08-03 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Anemia | 120 days
  Percentage of volunteers reaching normal Hb levels during the study.
Hemoglobin levels | 120 days
  Variation in hemoglobin levels (mg/dL)
Serum ferritin levels | 120 days
  Variation in serum ferritin levels (ug/l)

SECONDARY OUTCOMES:
Hemoglobin levels | 90 days
  Variation in hemoglobin levels (mg/dL)
Serum ferritin levels | 90 days
  Variation in serum ferritin levels (ug/l)
Body iron content | 120 days
  Variation in body iron content levels
Mean corpuscular volume | 120 days
  Variation in mean corpuscular volume (fL)
Red Blood Cell Distribution Width | 120 days
  Variation in Red Blood Cell Distribution Width (%)
Soluble transferrin receptor levels | 120 days
  Variation in soluble transferrin receptor levels (nmol/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Salud Global, Tumbes, Peru

REFERENCES:
- [Background] Suchdev PS, Jefferds MED, Ota E, da Silva Lopes K, De-Regil LM. Home fortification of foods with multiple micronutrient powders for health and nutrition in children under two years of age. Cochrane Database Syst Rev. 2020 Feb 28;2(2):CD008959. doi: 10.1002/14651858.CD008959.pub3. PMID 32107773
- [Background] Eichler K, Hess S, Twerenbold C, Sabatier M, Meier F, Wieser S. Health effects of micronutrient fortified dairy products and cereal food for children and adolescents: A systematic review. PLoS One. 2019 Jan 23;14(1):e0210899. doi: 10.1371/journal.pone.0210899. eCollection 2019. PMID 30673769
- [Background] Gera T, Sachdev HS, Boy E. Effect of iron-fortified foods on hematologic and biological outcomes: systematic review of randomized controlled trials. Am J Clin Nutr. 2012 Aug;96(2):309-24. doi: 10.3945/ajcn.111.031500. Epub 2012 Jul 3. PMID 22760566
- [Background] Finkelstein JL, Mehta S, Villalpando S, Mundo-Rosas V, Luna SV, Rahn M, Shamah-Levy T, Beebe SE, Haas JD. A Randomized Feeding Trial of Iron-Biofortified Beans on School Children in Mexico. Nutrients. 2019 Feb 12;11(2):381. doi: 10.3390/nu11020381. PMID 30759887
- [Derived] Alarcon-Yaquetto DE, Rueda-Torres L, Bailon N, Barreto PV, Malaga G. Accuracy of HemoCue301 portable hemoglobin analyzer for anemia screening in capillary blood from women of reproductive age in a deprived region of Northern Peru: An on-field study. PLoS One. 2023 Nov 14;18(11):e0293984. doi: 10.1371/journal.pone.0293984. eCollection 2023. PMID 37963155